CLINICAL TRIAL: NCT03438084
Title: The INTER-CARDIO Study: The Impact of Commonly Consumed Fat on Cardiovascular
Brief Title: The INTER-CARDIO Study: The Impact of Commonly Consumed Fat on Cardiovascular Health; a Randomised Controlled Trial
Acronym: INTER-CARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR-
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-08

CONDITIONS: Healthy Adults
Keywords: Interesterified; Postprandial; Lipid
MeSH Terms: interventions — Rapeseed Oil; Butter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interesterified (Experimental): Commercially available interesterifed fat spread. 50g fat.
  Interventions: Dietary Supplement: Interesterified fat
- Non- interesterified (Active Comparator): Commercially available non-interesterified fat. 50g fat.
  Interventions: Dietary Supplement: Non- interesterified fat
- Control (Active Comparator): Rapeseed oil. 50 g fat.
  Interventions: Dietary Supplement: Rapeseed oil
- Saturated fat control (Active Comparator): Butter. 50g fat
  Interventions: Dietary Supplement: Butter

INTERVENTIONS:
Dietary Supplement: Interesterified fat — 50 g fat provided as commercially available interesterified fat.
  Arms: Interesterified
Dietary Supplement: Non- interesterified fat — 50 g fat provided as commercially available non-interesterified fat.
  Arms: Non- interesterified
Dietary Supplement: Rapeseed oil — 50 g fat provided as commercially available rapeseed oil.
  Arms: Control
Dietary Supplement: Butter — 50g fat provided as commercially available spreadable butter
  Arms: Saturated fat control

SUMMARY:
The purpose of this study is to investigate whether there are differences in postprandial cardiometabolic metabolic indices following interesterified fats used commercially versus application appropriate non- interesterifed alternative fat.

DETAILED DESCRIPTION:
Aim: The current study aims to investigate the acute effects of commercially available interesterified fat versus versus application appropriate non- interesterifed alternative fat on 8 h postprandial cardiometabolic outcomes.

Hypothesis: Interesterified fat will induce a different cardiomtabolic response compared to a non interesterifed, application appropriate fat.

Subjects: Participants will include 40 healthy male and female volunteers aged between the ages of 35 and 75 years (since during this age metabolic changes start to take place).

Power calculation: Based on previous studies carried out by our group at King's College London, a sample size of 20 participants (males and females separately) will allow a 2.16% (percentage unit) difference in FMD to be detected (90% power, 0.05 alpha, SD 2.9. 50 participants will be recruited allowing for a 20% dropout rate.

Expected value:The study will provide novel information on the acute effects of commercially relevant processed fats on postprandial lipaemia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 35-75 years
* Healthy (free of diagnosed diseases listed in exclusion criteria)
* Able to understand the information sheet and willing to comply with study protocol
* Able to give informed consent

Exclusion Criteria:

* Medical history of myocardial infarction, angina, thrombosis, stroke, cancer, liver or bowel disease or diabetes
* Body mass index < 20 kg/m2 or > 35 kg/m2
* Plasma cholesterol ≥7.5 mmol/L
* Plasma triacylglycerol > 3 mmol/L
* Plasma glucose > 7 mmol/L
* Blood pressure ≥140/90 mmHg
* Current use of antihypertensive or lipid lowering medications
* Alcohol intake exceeding a moderate intake (> 28 units per week)
* Current cigarette smoker (or quit within the last 6 months)
* ≥ 20% 10-year risk of CVD as calculated using a risk calculator

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Up to 8 hours
  Flow mediated dilatation
Postprandial lipaemic response | Up to 8 hours
  Area under plasma TAG concentration/ time curve

SECONDARY OUTCOMES:
Postprandial lipaemic response | Up to 8 hours
  Postprandial plamsa total fatty acid composition and non esterifed fatty acid
Metabolomic for assessment of atherogenic potential (lipoprotein) analysis | Up to 8 hours
  Lipid concentrations and compositions of 14 lipoprotein subclasses, measured by NMR
Glycaemic response | Up to 8 hours
  Plasma glucose concentration
Insulinaemic response | Up to 8 hours
  Plasma insulin concnetration
Nitric oxide bioavailability | Up to 8 hours
  Plasma nitric oxide species and NADPH oxidase activity
Oxidative stress | Up to 8 hours
  Plasma 8-isoprostane F2a
Inflammatory response | Up to 8 hours
  Plasma IL-6

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Department of Nutritional Sciences, Faculty of Life Sciences and Medicine, Kings College London, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall WL, Alkoblan A, Gibson PS, D'Annibale M, Coekaerts A, Bauer M, Bruce JH, Lecomte B, Penhoat A, Laugerette F, Michalski MC, Salt LJ, Wilde PJ, Berry SE. Postprandial lipid and vascular responses following consumption of a commercially-relevant interesterified palmitic acid-rich spread in comparison to functionally-equivalent non-interesterified spread and spreadable butter: a randomised controlled trial in healthy adults. Food Funct. 2024 Mar 4;15(5):2733-2750. doi: 10.1039/d3fo05324e. PMID 38380649